CLINICAL TRIAL: NCT00812695
Title: Effects of Continuous Positive Airway Pressure in Patients With Resistant Hypertension and Obstructive Sleep Apnea
Brief Title: Effects of Continuous Positive Airway Pressure (CPAP) in Patients With Resistant Hypertension and Obstructive Sleep Apnea (OSA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Geraldo Lorenzi-Filho, MD; PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RH-OSA
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Obstructive Sleep Apnea; Refractory Hypertension
Keywords: Obstructive sleep apnea; Refractory hypertension; Heart remodeling; Arterial stiffness; CPAP
MeSH Terms: conditions — Sleep Apnea, Obstructive; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention)
- 2 (Active Comparator): CPAP
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Gold standard treatment for Obstructive sleep apnea
  Arms: 2

SUMMARY:
Obstructive sleep apnea (OSA) is an important cause of refractory hypertension but the impact of treatment with continuous positive airway pressure (CPAP) is not completely understood. The aim of this project is to study the effects of CPAP on blood pressure control and its influences on cardiac remodeling and arterial stiffness in patients with refractory hypertension and moderate or severe OSA.

DETAILED DESCRIPTION:
Study design Interventional, open-label, randomized.

Patients selection

Fifty refractory hypertensive patients with moderate-to-severe OSA, aged between 30 to 65 years old will be recruited from the outpatient clinics of the Heart Institute by the hospital staff.

Refractory hypertension will be defined as usually: blood pressure higher than or equal to 140x90 mmHg after a regimen of three drugs, including a diuretic for a minimum of 3 months. Initial evaluation will consist on ambulatory blood pressure measurement for 24 hours and a detailed clinical examination. Moderate to severe OSA will be defined as an apnea-hypopnea index > 15 evens per hour, after an overnight polysomnography.

Exclusion criteria include BMI >40 kg/m2; diabetes mellitus; aortic, heart and valve diseases; renal failure; other identifiable causes of hypertension, no adherence, use of cocaine, amphetamines, other illicit drugs, sympathomimetics (decongestants, anorectics), oral contraceptive hormones, nonsteroidal anti-inflammatory drugs.

Refractory hypertension Secondary causes of hypertension will be excluded using usual procedures from the Hypertension Unit.

Polysomnography All participants will be submitted to standard overnight polysomnography (EMBLA - Flagra hf. Medical Devices, Reykjavik, Iceland). The apnea-hypopnea index will be calculated as the total number of respiratory events (apneas plus hypopneas) per hour of sleep.

Apnea will be defined as an air flow cessation greater than 10 seconds and hypopnea as a reduction grater than 50% with oxygen saturation fall grater than 4% or arousal.

After recruitment, patients will be instructed about CPAP working by an experimented professional and another polysomnography will be done to adjust pressures. Hour counter will be used to check the adherence to CPAP.

Intervention Patients will be divided in two groups: medical treatment plus CPAP or medical treatment alone for 6 months without drug dose changing.

Twenty-four hour blood pressure monitoring Twenty-four hour blood pressure monitoring (system SpaceLabs 90207) will be used in all patients in the beginning and at the end of the study.

Arterial Stiffness Carotid-femoral arterial stiffness will be determined by Complior.

Echocardiography Echocardiography will be performed by using a commercially available machine.

ELIGIBILITY:
Inclusion Criteria:

* Refractory hypertensive patients with moderate-to-severe OSA, aged between 30 to 65 years old.

Exclusion Criteria:

* Aortic, heart and valve diseases
* Renal failure
* Other identifiable causes of hypertension, no adherence, use of cocaine, amphetamines, other illicit drugs, sympathomimetics (decongestants, anorectics), oral contraceptive hormones, nonsteroidal anti-inflammatory drugs.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Ambulatory blood pressure monitoring | Change from Baseline in Blood Pressure at 6 months

SECONDARY OUTCOMES:
Change from Baseline in Arterial stiffness at 6 months | baseline and 6 months
change from baseline in heart remodeling at 6 months | baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor), São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Pedrosa RP, Drager LF, de Paula LKG, Amaro ACS, Bortolotto LA, Lorenzi-Filho G. Effects of OSA treatment on BP in patients with resistant hypertension: a randomized trial. Chest. 2013 Nov;144(5):1487-1494. doi: 10.1378/chest.13-0085. PMID 23598607